CLINICAL TRIAL: NCT03633448
Title: An Open-label, Single-dose, Randomized, Two-way Crossover Study to Evaluate the Pharmacokinetics of Guaifenesin in Adults and Adolescents at Immediate-release Doses of 200 mg and 400 mg.
Brief Title: Study to Evaluate the Pharmacokinetics of Guaifenesin in Adults and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2011-GGE-06
Record Dates: First submitted 2018-08-14; First posted 2018-08-16 (Actual); Results first posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Mucinex® 1 x 200 mg (10 mL) (Experimental): 1 x 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate-release formulation
  Interventions: Drug: Children's Mucinex® Grape Flavor
- Mucinex® 1 x 400 mg (20 mL) (Experimental): 1 x 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate-release formulation
  Interventions: Drug: Children's Mucinex® Grape Flavor

INTERVENTIONS:
Drug: Children's Mucinex® Grape Flavor — 1 x 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate-release formulation
  Arms: Mucinex® 1 x 200 mg (10 mL)
Drug: Children's Mucinex® Grape Flavor — 1 x 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate-release formulation
  Arms: Mucinex® 1 x 400 mg (20 mL)

SUMMARY:
Evaluate the pharmacokinetics (PK), Safety and tolerability of guaifenesin (Mucinex®) in an immediate-release formulation when a single dose is administered in adolescents and in adults when compared to Children.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 12 and < 18 years of age or ≥ 18 and < 55 years of age.

   All females who were of childbearing potential had to be using one of the following acceptable birth control methods for the time periods specified:
   1. Intrauterine device (IUD) in place for at least 3 months prior to Day 1 of Period 1 through 30 days beyond study completion (Day 1 of Period 2).
   2. Barrier method (condom or diaphragm) with spermicide for at least 7 days prior to screening through 30 days beyond study completion (Day 1 of Period 2)
   3. Stable hormonal contraceptive (oral, depo injection, transdermal patch, or vaginal ring) for at least 3 months prior to Day 1 of Period 1 through 30 days beyond completion of study (Day 1 of Period 2).

   Note: Abstinence (sexually inactive) was not an acceptable form of contraception; however, abstinent female subjects could have been admitted to the study if they agreed, and had signed a statement to the effect, that upon becoming sexually active, would use a condom with spermicide from that time through 30 days beyond completion of the study (Day 1 of Period 2).

   Females ≥ 18 years of age of non-childbearing potential must have been surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to Day 1 of Period 1 or hysterectomy and/or bilateral oophorectomy at least 3 months prior to Day 1 of Period 1) or post-menopausal ≥ 2 years prior to Day 1 of Period 1. A follicle stimulating hormone (FSH) level > 40 miU/mL must have been obtained and in the record for any post-menopausal female experiencing their last menses < 2 years prior to Day 1 of Period 1.
2. Negative urine pregnancy test at Screening and each Check-in for all female subjects.
3. Good general health as determined by the PI's review of medical history, physical examination, vital sign measurements (after 2 minutes resting in the seated position), and clinical laboratory measures.
4. For subjects ≥ 18 and < 55 years of age, body mass index (BMI) of 19 to 29 kg/m2, inclusive. (BMI = weight (kg)/[height (m)]2).
5. Subjects ≥ 12 and < 18 years of age had to be > 5th percentile and less than the 95th percentile for weight and BMI of ≥ 18 to ≤ 28 kg/m2 based on age and gender.
6. Non-tobacco users, who had not used nicotine or nicotine-containing products for at least 1 year prior to Day 1 of Period 1.
7. Negative finding on tests for hepatitis B surface antigen (HBsAG), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV).
8. Negative urine screen for drugs of abuse and alcohol at Screening and each Check-in.
9. Likely to be compliant and complete the study, and if < 18 years of age had parent(s) or legally authorized representative(s) likely to be compliant with study requirements, according to the PI.
10. Able to read, understand, and sign the informed consent, after the nature of the study had been explained, and had read, signed, and dated an IRB-approved informed consent/assent form for subjects to participate in the study. Additionally, for subjects < 18 years of age, a parent(s) or legally authorized representative(s), had to read, sign, and date an IRB-approved informed consent/assent form for subjects < 18 years of age to participate in the study.
11. Subjects < 18 years of age must have met the following at-risk requirements:

    1. Frequency - a history of frequent upper respiratory infections (URIs) defined as > 4 infections per year for adolescents aged ≥ 12 to < 18 yrs, AND;
    2. Exposure - Another family member in the home who was ill with URI/common cold or a child in the family who was attending preschool or school with ≥ 6 children in the group, AND;
    3. Crowding - Greater than (>) 4 persons living in the home or > 3 persons sleeping in one bedroom.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical examination, vital sign measurements, ECG findings, or clinical laboratory findings (as determined by the PI), including a hemoglobin value < 12 gm/dL at Screening.
2. Females who were pregnant or nursing.
3. History of hypersensitivity reaction to guaifenesin or to EMLA® cream (eutectic mixture of local anesthetic) or its components (lidocaine + prilocaine as local anesthetic).
4. Receipt of an investigational drug within 30 days prior to Day 1 of Period 1.
5. Abnormal diet (for whatever reason) during the 30 days prior to Day 1 of Period 1.
6. Donation of blood or significant loss of blood within 56 days prior to Day 1 of Period 1.
7. Donation of plasma within 14 days prior to Day 1 of Period 1.
8. Known or suspected use of illicit drugs (i.e., opiates, barbiturates, marijuana, et. al.).
9. The use of any medication on a chronic basis, with the exception of hormonal contraceptives for women of child-bearing potential. An appropriate drug free period for prescription or OTC drugs should have been provided to wash out any especially long half-life drugs.
10. Alcoholism or medicinal product or drug abuse within the past two years or excessive alcohol consumption (more than 10 units per week) (one unit was defined as 5 ounces of wine, 12 ounces of beer, or 1.5 ounces of spirits (i.e., "hard" liquor such as gin, whiskey, or vodka, et. al.). The subject was not to experience tolerance, withdrawal, compulsive use, or substance related problems such as medical complications, disruption in social and family relationships, vocational or financial difficulties, or legal problems.
11. Consumption of grapefruit, pummelo, Seville orange or grapefruit juice within 14 days prior to dosing with study medication. Subjects had to be willing to abstain from consuming any of these products during the study.
12. Related to persons involved directly or indirectly with the conduct of this study (i.e., PI, Sub-Investigators, Study Coordinators, other study personnel, employees of Reckitt Benckiser, and the families of each).

Subject Exclusion Criteria at Check-In

1. Any significant change from Screening in medical history, medication history, alcohol consumption, or tobacco/nicotine use, in the opinion of the PI.
2. Reports any known enzyme-inducer, enzyme-inhibitor, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides since Screening, unless approved by Reckitt Benckiser.
3. Reports any other prescription or OTC drug or herbal remedy since Screening (except for low-dose contraceptives, multivitamins, and/or fluoride supplements) unless allowed by Reckitt Benckiser.
4. If female, a positive urine pregnancy test.
5. Had an acute illness since Screening, unless allowed by Reckitt Benckiser.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-06-18 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: Total 24 subjects were enrolled in the study and all 24 completed the study.
Groups:
- 200mg Dose of Guaifenesin, Then 400mg Dose of Guaifenesin: Treatment Sequences 1 [6 adolescents/6 adults]: Treatment A in Period 1, then Treatment B in Period 2
  Treatment A: Single 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  Treatment B: Single 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  There was a 7 days washout period between each administration.
- 400mg Dose of Guaifenesin, Then 200mg Dose of Guaifenesin: Treatment Sequences 2 [6 adolescents/6 adults]: Treatment B in Period 1, then Treatment A in Period 2.
  Treatment B: Single 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  Treatment A: Single 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  There was a 7 days washout period between each administration.
Period: Period 1 (1 Day)
Arm/Group | 200mg Dose of Guaifenesin, Then 400mg Dose of Guaifenesin | 400mg Dose of Guaifenesin, Then 200mg Dose of Guaifenesin
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout (7 Days)
Arm/Group | 200mg Dose of Guaifenesin, Then 400mg Dose of Guaifenesin | 400mg Dose of Guaifenesin, Then 200mg Dose of Guaifenesin
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2 (1 Day)
Arm/Group | 200mg Dose of Guaifenesin, Then 400mg Dose of Guaifenesin | 400mg Dose of Guaifenesin, Then 200mg Dose of Guaifenesin
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Adolescent; Adult: Treatment A: Single 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  Treatment B: Single 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
  There was a 7 days washout period between each administration.
- Total: Total of all reporting groups
Arm/Group | Adolescent | Adult | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.3 (1.71) | 32.2 (12.42) | 23.2 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 5 | 4 | 9
Race [Count of Participants; unit: Participants]
  Asian | 1 | 2 | 3
  Black or African American | 10 | 8 | 18
  White | 1 | 2 | 3
Ethnicity [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Non-Hispanic and Non-Latino | 11 | 12 | 23
Height [Mean (Standard Deviation); unit: cm] | 163.9 (7.69) | 166.83 (10.954) | 165.35 (9.379)
Weight [Mean (Standard Deviation); unit: kg] | 56.03 (7.198) | 66.88 (11.611) | 61.45 (10.955)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 20.78 (1.482) | 23.98 (3.168) | 22.38 (2.917)

OUTCOME MEASURES:

1. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC(0-t)) of Guaifenesin
Description: Area under the plasma concentration versus time curve from time 0 to the time of the last measurable concentration, as calculated by the linear trapezoidal method.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: Pharmacokinetic (PK) Data Sets included only those subjects who swallowed the whole dose (did not spit it out), did not vomit within one hour of dosing, and who had a sufficient number of plasma concentrations to estimate the primary PK parameters for at least one dose level.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Groups:
- Treatment A (Adolescents); Treatment A (Adults): Treatment A: Single 200 mg (10 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
- Treatment B (Adolescents); Treatment B (Adults): Treatment B: Single 400 mg (20 mL) Children's Mucinex® Grape Flavor 100 mg Guaifenesin/5 mL immediate Release by oral syringe under overnight fast.
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng*hr/mL | 1990 (929) | 1700 (742) | 4390 (1590) | 3910 (1500)

2. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to Infinity (AUC(0-inf)) of Guaifenesin
Description: Area under the plasma concentration versus time curve from time 0 to infinity, calculated as AUC 0-t + C last/kel, where C last is the last measurable concentration and kel is the apparent first-order terminal elimination rate constant.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng*hr/mL | 2090 (916) | 1710 (744) | 4400 (1600) | 3930 (1500)

3. Primary Outcome: Percent of AUC 0-inf Extrapolated (AUC%Extrapolated)
Description: Percent of AUC 0-inf extrapolated, calculated as (1 - AUC 0-t / AUC 0-inf) x 100.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Percentage | 0.469 (0.426) | 0.736 (0.775) | 0.476 (0.431) | 0.386 (0.134)

4. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Pharmacokinetic Parameter (Cmax) Maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
ng/mL | 1360 (968) | 887 (419) | 2690 (1220) | 1950 (739)

5. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Guaifenesin
Description: Pharmacokinetic Parameter (Tmax) Time of the maximum observed plasma concentration.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr | 0.458 (0.209) | 0.711 (0.403) | 0.524 (0.325) | 0.646 (0.345)

6. Primary Outcome: Apparent First-order Terminal Elimination Half-life (t½)
Description: Apparent first-order terminal elimination half-life, calculated as ln(2)/kel.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr | 1.05 (0.173) | 1.10 (0.228) | 0.963 (0.129) | 0.963 (0.0899)

7. Primary Outcome: Apparent First-order Terminal Elimination Rate Constant (Kel)
Description: Apparent first-order terminal elimination rate constant calculated from a semilog plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares (LS) regression analysis using the maximum number of points (e.g., three or more non-zero plasma concentrations) in the terminal log-linear phase.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, and 8 hours
Population: PK Data Sets
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
1/hr | 0.678 (0.100) | 0.655 (0.122) | 0.731 (0.0928) | 0.726 (0.0757)

8. Secondary Outcome: Number of Adverse Events (AEs) of Participants
Description: Intensity determination:
  Mild=AE does not limit usual activities;subject may experience slight discomfort; Moderate= AE results in some limitation of usual activities; subject may experience significant discomfort; Severe=AE results in an inability to carry out usual activities; subject may experience intolerable discomfort or pain; Unlikely=Slight but remote chance that the AE was caused by study drug but the balance of judgment is that it was most likely not due to the study drug Possible=Reasonable suspicion that the AE was caused by the study drug; Probable=Most likely that the AE was caused by study drug.
Time Frame: Upto Day 1
Population: PK Data Sets
Measure: Number; unit: Events
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
Number analyzed (Participants) | 12 | 12 | 12 | 12
Events
  TEAE by severity: Mild | 0 | 0 | 0 | 1
  TEAE by severity: Moderate | 0 | 0 | 0 | 1
  TEAE by severity: Severe | 0 | 0 | 0 | 0
  Relationship to Drug: Definite | 0 | 0 | 0 | 0
  Relationship to Drug: Probable | 0 | 0 | 0 | 0
  Relationship to Drug: Possible | 0 | 0 | 0 | 0
  Relationship to Drug: Unlikely | 0 | 0 | 0 | 0
  Relationship to Drug: None | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to Day 14
Arm/Group | Treatment A (Adolescents) | Treatment A (Adults) | Treatment B (Adolescents) | Treatment B (Adults)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (Adolescents) (N=12) | Treatment A (Adults) (N=12) | Treatment B (Adolescents) (N=12) | Treatment B (Adults) (N=12)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No